CLINICAL TRIAL: NCT06613230
Title: Improved Early Diagnosis and Survival in Female Pelvic Cancer (e.g. Ovarian Cancer) With OC Detect, (Pilot Study)
Brief Title: Improved Early Diagnosis in Female Pelvic Cancer With OC Detect
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Linkoeping University (Other Government); VOC Diagnostics (Industry)
Responsible Party: Principal Investigator, Christer Borgfeldt, Professor in Obsterics and Gynaecology at Lund University, Region Skane
Other Study IDs: 232100-0255; VOC-CLIN-001 (Other: VOC Diagnostics)
Record Dates: First submitted 2024-08-26; First posted 2024-09-25 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Breast Cancer; Lymphoma; Malignant Melanoma; Sarcoma
Keywords: in vitro diagnostic; volatile organic compound, VOC; electronic nose; blood plasma samples; cancer diagnosis
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Breast Neoplasms; Lymphoma; Melanoma; Sarcoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cancer: Blood plasma samples from female patients with ovarian cancer of stage I-IV or borderline tumours, stored in biobanks in Sweden.
  Also blood samples from female patients with other cancer types (endometrial, lymphoma, breast, malignant melanoma and sarcoma)
- Healthy blood donors: Healthy blood donors samples from women aged 18-70 years

SUMMARY:
The goal of this observational study is to learn if so called Volatile Organic Compounds (VOCs) in blood can be used for early diagnosis of ovarian cancer. The main question it aims to answer is:

Can OC Detect, a new in vitro diagnostic instrument, distinguish between VOC patterns in blood plasma from women with ovarian cancer (especially in early stage) and VOC patterns in helthy women? Participants are previosuly diagnosed patients with ovarian cancer, who agreed to store their blood samples in biobanks for future medical research purposes. Healthy female blood donors serve as benign control blood samples.

DETAILED DESCRIPTION:
Pelvic Endometrial and Ovarian cancer (ovarian-/tubal-/peritoneal cancer) is the sixth and seventh most frequent type of cancer and ovarian cancer the fourth leading cause of cancer related death among Swedish women. Endometrial cancer gives mostly early symptoms but two thirds of patients with ovarian cancer are diagnosed with advanced stage of the disease, and this is reflected in poor outcome. Early diagnosis is challenging especially in ovarian cancer.

Plasma protein biomarker panels with improved diagnostic performance and predicting survival in patients with ovarian tumors have been performed by several research groups. The sensitivity is good, but specificity is today not good enough for screening purposes. Several blood-based protein biomarker candidates for endometrial cancer detection have been reported but the protein biomarkers have so far only clinical relevance in advanced or recurrent endometrial cancers. However, there is a need for improved more specific broader biomarker panels for discrimination between localized or metastatic disease and preoperative risk stratification especially in endometrial cancer patients. Such improved biomarker panels would be able to predict metastatic disease and guide adjuvant chemotherapy treatment.

Endogenous volatile organic compounds (VOCs) are products of metabolic activity in the body and changes to these VOCs can be characteristic of specific disease processes such as cancer development. Analyses in plasma of VOCs such as triethylamine, pyridine, toluene, etc. with Field-Effect-Transistor (FET) -based gas sensors have shown to be able to measure VOCs very accurately in low concentrations (Bastuck thesis, 2009). The metabolism in cancer cells vastly differs from that of healthy cells. Elevated glycolysis leads to increases in lactate and fumarate metabolites resulting in altered VOC abundances in exhaled breath. Experimental data indicate that the detection of VOCs released by various cancer cells may be useful in early diagnoses of cancer. In patients with ovarian cancer, analyzes of specific VOC: s in blood has shown promising results to discriminate patient with ovarian cancer from healthy women (Horvath). The investigators have very recently in 37 patients out 38 with ovarian cancer found VOC indicating cancer which indicates a preliminary sensitivity of 97 %. In the total material of 68 analyzed samples, 3 false positive results were found which indicates a specificity of 90 %. In a population with 1 % malignancy the positive predictive value would be almost 10 % and negative predictive value 99.9 %.

In the current study, samples from more ovarian cancer patients will be included, and also samples from patients with other cancer types (totally 245 patients, of which 50 ovarian cancers). The aim will be to see if good sensitivity and specificity can be achived with larger patient population (same or better values than in the previous study). Special focus will be put on early stages of ovarian cancer, as well as borderline tumours. The investigators aim also to see how distinct is VOC pattern for ovarian cancer compared to the VOC patterns for the other cancer forms. Finally, the study will give preliminary answer if VOC patterns for the other types of cancer (i.e., breast, colorectal, bladder, endometrie, cervix, ...) is specific so it could be used in the future for development of dedicated diagnostic tools for those diseases.

ELIGIBILITY:
Inclusion Criteria:

* Blood plasma (1ml) from patients with ovarian cancer or borderline ovarian tumors, or other cancer tumors (endometrial, lymphoma, breast, malignant melanoma, sarcoma)
* Blood plasma (1 ml) from healthy volunteer controls
* Signed informed consent by cancer patients for use of biobank blood samples in research
* Signed informed consent by healthy blood donors for use in research

Exclusion Criteria:

* < 18 years (both for cancer patients and healthy blood donors)
* Man (healthy blood donors)
* >70 years (healthy blood donors)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood plasma samples from patients with ovarian and other types of cancer admitted to cancer clinics in south part of Sweden (Region Skane), who are diagnbosed with cancer and who have signed informed consent for storing of their blood samples in biobanks for future reseatrch purposes. The patients are psudo-anonymous.
  Healthy blood donors from Linköping University hospital who have signed informed consent allowing use of their blood in research after local approval. The helthy donors are anonymous.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of VOC algorithm for ovarian cancer diagnosis | From time of blood sample collection for cancer diagnosis until the time of VOC measurement, assessed 1 year - 15 years post diagnosis
  Classification of features of the VOC patterns in plasma of each ovarian cancer patient and each healthy control as cancer or healthy control, by OC Detect algorithm. Determination of false positives (FP)/ false negative (FN)/ true positive (TP)/ true negative (TN) diagnoses based on comparison to the ground truth clinical diagnoses from biobank and healthy controls. Determination of sensitivity, specificity and accuracy.

SECONDARY OUTCOMES:
Performance of VOC algorithm for other patients with endometrial, breast, lymphoma, malignant melanoma and sarcoma patients. | From time of blood sample collection for cancer diagnosis until the time of VOC measurement, assessed 1 year - 15 years post diagnosis
  Classification of features of the VOC patterns in plasma of each cancer patient and each healthy control as cancer or healthy control, by OC Detect algorithm. Determination of false positives (FP)/ false negative (FN)/ true positive (TP)/ true negative (TN) diagnoses based on comparison to the ground truth clinical diagnoses from biobank and healthy controls. Determination of sensitivity, specificity and accuracy for each cancer type.
Preliminary performance for an algorithm for all cancer types in the study, with special attention to ovarian cancer compared to the other cancer types | From time of blood sample collection for cancer diagnosis until the time of VOC measurement, assessed 1 year - 15 years post diagnosis
  Classification of features for VOC patterns in plasma of all cancer types as specific other cancer type or as healthy control, after training of new algorithm for discrimination all cancer types in this study (multiple classification).

OTHER OUTCOMES:
Performance of VOC algorithm for ovarian cancer diagnosis on cancer stage level | From time of blood sample collection for cancer diagnosis until the time of VOC measurement, assessed 1 year - 15 years post diagnosis
  Classification of features of the VOC patterns in plasma of each ovarain cancer patient and each healthy control as ovarain cancer stage (borderline - stage I-II or stage III-IV) or healthy control, by OC Detect algorithm. Determination of preliminary sensitivity, specificity and accuracy for each cancer stage.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eriksson, Ass Prof, Study Director — Linkoeping University
Locations (2):
- Sweden (2):
  - Linkoping University, Linköping
  - Region Skane, Lund

IPD SHARING:
Plan to Share IPD: No